CLINICAL TRIAL: NCT07096973
Title: Cardiac REhabilitation COhort at the Medicine Campus DaVos to invEstigate Recovery
Acronym: RECOVER
Status: Recruiting | Type: Observational
Sponsor: Hochgebirgsklinik Davos (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02560
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Rehabilitation; Heart Failure; Cardiac Arrest (CA); ACS (Acute Coronary Syndrome); CABG; Valve Anomalies; LVAD (Left Ventricular Assist Device); Heart Transplantation; Arrhythmia
Keywords: cardiovascular diseases; cardiac rehabilitation
MeSH Terms: conditions — Heart Failure; Heart Arrest; Acute Coronary Syndrome; Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Blood (EDTA-blood, serum, plasma (EDTA), citrated), DNA, RNA, washed erythrocytes, PBMCs (peripheral blood mononuclear cell)
  * Urine
  * Stool
  * Tissue/ cells
  * Saliva
  * Hair
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RECOVER study, titled Cardiac Rehabilitation Cohort at the Medicine Campus Davos for Exploration of Recovery, is a prospective, non-interventional, monocentric cohort study conducted at the Hochgebirgsklinik Davos. The study is sponsored by Medicine Campus Davos AG and the Kühne Foundation, with an estimated start date in July 2025 and planned completion by December 2034, with the possibility of extension.

The principal investigator of the study is PD Dr. David Niederseer from Hochgebirgsklinik Davos, who also represents the study. The research team includes co-investigators such as Prof. Dr. Stefan Blankenberg and Prof. Dr. Andreas Ziegler from Cardio-CARE, Medicine Campus Davos, as well as Dr. Jan Vontobel from Hochgebirgsklinik Davos.

The study will enroll patients referred to Hochgebirgsklinik Davos for cardiac rehabilitation who provide informed consent. Cardiac rehabilitation is an evidence-based therapy for patients with heart disease, including those who have undergone cardiac procedures or surgeries.

The primary objectives are to evaluate baseline patient characteristics, rehabilitation strategies, predictors of recovery, and clinical outcomes during and after rehabilitation. To support this, a detailed database and biobank will be established to allow for comprehensive phenotyping, extensive clinical assessments, and long-term follow-up.

RECOVER seeks to gain translational insights into how patient-specific factors - such as genetics, plasma, digital and clinical biomarkers, and comorbidities - influence long-term clinical outcomes. The goal is to identify modifiable risk factors to optimize individualized therapeutic approaches in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CR at the HGK
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Insufficient knowledge of the German language to understand study documents, the interview, or questionnaires interview without translation
* Physical or psychological incapability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to HGK for inpatient CR will be screened for eligibility according to inclusion and exclusion criteria. Study inclusion requires written informed consent, and the study and all -related procedures will be performed according to the Declaration of Helsinki. The study plans to enroll approximately 1'000 patients per year.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2035-08-05 (Estimated); Study Completion 2040-08-05 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular mortality, non-fatal myocardial infarction, non-fatal stroke, and hospitalization for heart failure | Follow-up 1, 5 and 10 years after inclusion
  Outcome assessment will be conducted through a combination of structured telephone follow-up, systematic collection of relevant medical records from the time of inclusion to the follow-up visit, patient-completed questionnaires, and analysis of data from national health and mortality registries.
Incidence of all-cause rehospitalization post cardiac intervention or surgery | Follow-up 1, 5 and 10 years after inclusion
  All-cause rehospitalization is defined as any unplanned hospital admission, regardless of cause, occurring following the index cardiac intervention or surgery. This includes admissions to any inpatient care facility for diagnostic, therapeutic, or emergency reasons, excluding planned elective procedures or routine follow-up admissions. Data will be obtained through structured follow-up, review of relevant hospital records, and linkage with national health insurance and hospital discharge registries to ensure comprehensive capture of rehospitalization events.

SECONDARY OUTCOMES:
Patient reported quality of life (QoL) | Follow-up 1, 5 and 10 years after inclusion
  Quality of life will be assessed using the EuroQol 5-Dimension (EQ-5D) questionnaire, a validated patient-reported outcome measure, administered at baseline and follow-up. The EQ-5D index score ranges from less than 0 (indicating health states worse than death) to 1 (perfect health), with higher scores reflecting better health-related quality of life. Changes in index scores will be analyzed to evaluate the effects of cardiac rehabilitation.
Re-surgery / Re-intervention | Follow-up 1, 5 and 10 years after inclusion
  The incidence of repeat cardiovascular surgery or catheter-based interventions will be recorded within the follow-up period. This includes any planned or unplanned procedures related to the index condition (e.g., valve re-surgery, revascularization) and will be verified through medical records and registry linkage.
New-Onset Atrial Fibrillation | Follow-up 1, 5 and 10 years after inclusion
  New-onset atrial fibrillation is defined as a first documented episode of AF after the index cardiac intervention or surgery, verified by ECG or rhythm monitoring. Occurrence will be assessed through medical records, telemetry data, and clinical follow-up.
Cognitive Function | Follow-up 1, 5 and 10 years after inclusion
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a standardized screening tool that evaluates multiple cognitive domains including memory, attention, executive function, and processing speed. Scores range from 0 to 30, with higher scores indicating better cognitive performance. Assessments will be conducted at baseline and follow-up to detect changes or cognitive decline following the intervention.
Functional Capacity | Follow-up 1, 5 and 10 years after inclusion
  Functional capacity will be objectively assessed at baseline and discharge using the standardized 6-minute walk test (6MWT). At follow-up, functional status will be evaluated through patient-reported outcomes collected via structured interviews and questionnaires to estimate changes in physical performance and exercise tolerance over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hochgebirgsklinik Davos, Davos, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No